CLINICAL TRIAL: NCT04389671
Title: A Multicenter, Single-Treatment Study to Assess the Safety and Tolerability of Lyophilized Lucinactant in Adults With COVID-19 Associated Acute Lung Injury
Brief Title: The Safety and Preliminary Tolerability of Lyophilized Lucinactant in Adults With Coronavirus Disease 2019 (COVID-19)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Windtree Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-CL-2001a
Record Dates: First submitted 2020-05-13; First posted 2020-05-15 (Actual); Results first posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: COVID-19; Acute Lung Injury/Acute Respiratory Distress Syndrome (ARDS)
MeSH Terms: conditions — COVID-19; Acute Lung Injury; Respiratory Distress Syndrome | interventions — lucinactant; sinapultide; Surface-Active Agents

STUDY DESIGN:
Intervention Model Description: Open-label, single treatment of reconstituted Lucinactant, delivered as an intratracheal liquid.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lyophilized Lucinactant (Experimental): Lyophilized Lucinactant reconstituted with sterile water for injection
  Interventions: Drug: Lucinactant

INTERVENTIONS:
Drug: Lucinactant — Lucinactant administered as a liquid at a dose of 80 mg total phospholipids (TPL)/kg lean body weight delivered
  Other Names: Sinapultide (KL4) Surfactant

SUMMARY:
This is a multicenter, single-treatment study. Subjects will consist of adults with COVID-19 associated acute lung injury who are being cared for in a critical care environment.

DETAILED DESCRIPTION:
This is a multicenter, single-treatment study. Subjects will consist of adults with COVID-19 associated acute lung injury who are being cared for in a critical care environment.

Lucinactant is a synthetic surfactant that, in its liquid form (SURFAXIN®), is approved by the United States Food and Drug Administration (NDA 021746) for the prevention of respiratory distress syndrome (RDS) in premature infants at high risk for RDS.

It has been studied in over 2000 children and adults. Preliminary data from animal and adult human studies indicate that lucinactant may be able to benefit those with acute respiratory distress syndrome (ARDS) in the context of COVID-19 infection, improving oxygenation and lung compliance. When given to intubated patients, Lucinactant could potentially decrease the duration of ventilation.

Lucinactant has an extensive safety profile in different patient populations for different indications.

It is hypothesized that lucinactant may improve the respiratory status of patients suffering from COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form (ICF) by the subject or legally authorized representative;
* Age 18-75 (inclusive);
* Assay positive for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) virus, preferably by polymerase chain reaction (PCR);
* Endotracheal intubation and mechanical ventilation (MV), within 7 days of initial intubation;
* In-dwelling arterial line;
* PaO2/FiO2 (P/F) ratio < 300;
* Mean blood pressure ≥ 65 mmHg, immediately before enrollment;
* Bilateral infiltrates seen on frontal chest radiograph.

Exclusion Criteria:

* Life expectancy < 48 hours or do not resuscitate orders;
* Severe lung disease (home O2, forced expiratory volume at one second [FEV1] < 2 liters) not likely to respond to therapy or profound hypoxemia (ie, oxygen index [OI] ≥ 25 or P/F ratio < 100);
* Severe renal impairment (creatinine clearance < 30 mL/min);
* Within the last 6 months has received, or is currently receiving, immunosuppression therapy (azathioprine, cyclophosphamide or methotrexate) or any transplant recipient;
* Clinically significant cardiac disease that adversely effects cardiopulmonary function:

  1. Acute coronary syndromes or active ischemic heart disease (as assessed by the PI using troponin and ECG)
  2. Cardiac ejection fraction < 40% (if known);
  3. Need for multiple-dose vasopressors to support blood pressure (single dose vasopressors, such as Levophed™ ≤ 0.1 mcg/kg/min are allowed);
  4. Cardiogenic pulmonary edema as the etiology of the current respiratory distress;
  5. Evidence of myocarditis or pericarditis;
* Neuromuscular disease;
* Neutropenia (ANC < 1000);
* Active malignancy that impacts treatment decisions or life expectancy related to the trial;
* Suspected concomitant bacterial or other viral lung infection. Bacterial infection defined as white blood count (WBC) > 15k and positive blood/urine/sputum culture results within 72 hours.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuh-Chin T Huang, MD, MHS, Principal Investigator — Duke University; Steve G Simonson, MD, Study Director — Windtree Therapeutics
Locations (11):
- United States (7):
  - University California San Diego - Jacobs Medical Center, La Jolla, California
  - University of California San Diego - Medical Center, Hillcrest, San Diego, California
  - Augusta University Health, Augusta, Georgia
  - University of Kentucky, Lexington, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
- Argentina (4):
  - Fundacion Sanatorio Güemes, Buenos Aires
  - Hospital Alemán, Buenos Aires
  - Hospital Italiano de Bueno Aires, Buenos Aires
  - CEMIC - Centro de Educacion Medica e Investigaciones Clinicals, Buenos Aires

IPD SHARING:
Plan to Share IPD: No
The preparation and submittal for publication of a manuscript containing the study results shall be in accordance with a process determined by a mutual written agreement among Windtree and participating institutions.
  The publication or presentation of any study results shall comply with all applicable privacy laws, including but not limited to HIPAA. This trial will be registered at ClinicalTrials.gov, and results information from this trial will be submitted. In addition, every attempt will be made to publish results in peer-reviewed journals.

REFERENCES:
- [Derived] Lee CK, Merriam LT, Pearson JC, Lipnick MS, McKleroy W, Kim EY. Treating COVID-19: Evolving approaches to evidence in a pandemic. Cell Rep Med. 2022 Feb 9;3(3):100533. doi: 10.1016/j.xcrm.2022.100533. eCollection 2022 Mar 15. PMID 35474746
- [Derived] Cohen CL, Walker KH, Hsiang M, Sonenthal PD, Riviello ED, Rouhani SA, Lipnick MS, Merriam LT, Kim EY. Combating information chaos: a case for collaborative clinical guidelines in a pandemic. Cell Rep Med. 2021 Aug 17;2(8):100375. doi: 10.1016/j.xcrm.2021.100375. Epub 2021 Jul 27. PMID 34337553

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant enrolled: 05 January 2021 Last participant completed: 20 February 2022 Enrollment occurred in hospital
Pre-assignment Details: No wash-out or run-in
Period: Overall Study
Arm/Group | Lyophilized Lucinactant
Started | 20
Completed | 13
Not Completed | 7
Not completed — Death | 7

BASELINE CHARACTERISTICS:
Population: One enrolled participant did not receive study treatment
Arm/Group | Lyophilized Lucinactant
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (13.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 11
  More than one race | 2
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Argentina | 2
  United States | 17
Oxygen Index [Mean (Standard Deviation); unit: index] — OI is an index value, calculated as the fraction of inspired oxygen (FiO2) times mean airway pressure (Paw) divided by the partial pressure of oxygen in the artery (PaO2).
  It is a calculation that measures the fraction of inspired oxygen and its usage within the body, and a lower value is better. Values can range from 0 to 1000; values under 25 are correspond with a good outcome.
  index | 10.7 (6.17)

OUTCOME MEASURES:

1. Primary Outcome: Oxygen Index (OI)
Description: Change from baseline in OI. OI is an index value, calculated as (Mean Airway Pressure [Paw]) x (Fraction of Inspired Oxygen [FiO2]) x (100) / (Partial Pressure of Oxygen [PaO2]) measured using mean and standard deviation.
  It is a calculation that measures the fraction of inspired oxygen and its usage within the body, and a lower value is better. Values can range from 0 to 1000; values under 25 are correspond with a good outcome.
Time Frame: Baseline through 12 hours post initiation of dosing
Population: All participants that received study medication
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Lyophilized Lucinactant
Number analyzed (Participants) | 19
index | -0.91 (3.14)

2. Secondary Outcome: Fraction of Inspired Oxygen (FiO2)
Description: Change from baseline in FiO2 measured using mean and standard deviation. FiO2 level, ranging from 0.21 (room air) to 1.00 (i.e., 21% to 100%)
Time Frame: Baseline through 24 hours post initiation of dosing
Population: All participants that received study medication
Measure: Mean (Standard Deviation); unit: fraction of oxygen
Arm/Group | Lyophilized Lucinactant
Number analyzed (Participants) | 19
fraction of oxygen | -0.05 (0.230)

3. Secondary Outcome: Partial Pressure of Oxygen (PaO2)
Description: Change from baseline in PaO2 measured using mean and standard deviation
Time Frame: Baseline through 24 hours post initiation of dosing
Population: All participants that received study medication
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lyophilized Lucinactant
Number analyzed (Participants) | 19
mmHg | -2.0 (27.63)

4. Secondary Outcome: Oxygenation From Pulse Oximetry (SpO2)
Description: Change from baseline in SpO2 measured using mean and standard deviation
Time Frame: Baseline through 24 hours post initiation of dosing
Population: All participants that received study medication
Measure: Mean (Standard Deviation); unit: percent of blood oxygen saturation
Arm/Group | Lyophilized Lucinactant
Number analyzed (Participants) | 19
percent of blood oxygen saturation | -0.4 (4.36)

5. Secondary Outcome: Oxygen Index (OI)
Description: Change from baseline in OI. OI is an index value, calculated as Paw x FiO2 x 100 / PaO2, measured using mean and standard deviation.
  It is a calculation that measures the fraction of inspired oxygen and its usage within the body, and a lower value is better. Values can range from 0 to 1000; values under 25 are correspond with a good outcome.
Time Frame: Baseline through 24 hours post initiation of dosing
Population: All participants that received study medication
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Lyophilized Lucinactant
Number analyzed (Participants) | 19
index | -1.46 (5.328)

6. Secondary Outcome: Partial Pressure of Carbon Dioxide (PaCO2)
Description: Change from baseline in PaCO2 measured using mean and standard deviation
Time Frame: Baseline through 24 hours post initiation of dosing
Population: All participants that received study medication
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lyophilized Lucinactant
Number analyzed (Participants) | 19
mmHg | -3.6 (10.37)

7. Secondary Outcome: End Tidal Carbon Dioxide (ETCO2)
Description: Change from baseline in ETCO2 measured using mean and standard deviation
Time Frame: Baseline through 24 hours post initiation of dosing
Population: All participants that received study medication
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lyophilized Lucinactant
Number analyzed (Participants) | 19
mmHg | -1.6 (4.88)

8. Secondary Outcome: PaO2 to FiO2 (P/F) Ratio
Description: Change from baseline in ratio of arterial oxygen concentration to fraction of inspired oxygen (P/F ratio) and/or ratio of pulse oximetric saturation to fraction of inspired oxygen (P/F and/or S/F ratios) measured using mean and standard deviation.
Time Frame: Baseline through 24 hours post initiation of dosing
Population: All participants that received study medication
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Lyophilized Lucinactant
Number analyzed (Participants) | 19
ratio | -3.87 (71.26)

9. Secondary Outcome: SpO2 to FiO2 (S/F) Ratio
Description: Change from baseline in ratio of pulse oximetric saturation to fraction of inspired oxygen (S/F ratio) measured using mean and standard deviation.
Time Frame: Through 24 hours
Population: All participants that received study medication
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Lyophilized Lucinactant
Number analyzed (Participants) | 19
ratio | 15.35 (65.32)

10. Secondary Outcome: Plateau Pressure (PPLAT)
Description: Change from baseline in PPLAT, as measured on the ventilator, measured using mean and standard deviation.
Time Frame: Through 24 Hours
Population: All participants that received study medication
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | Lyophilized Lucinactant
Number analyzed (Participants) | 19
cm H2O | 0.5 (3.36)

11. Secondary Outcome: Peak Inspiratory Pressure (PIP)
Description: Change from baseline in PIP, as measured on the ventilator, measured using mean and standard deviation.
Time Frame: Baseline through 24 hours post initiation of dosing
Population: All participants that received study medication
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | Lyophilized Lucinactant
Number analyzed (Participants) | 19
cm H2O | -1.0 (4.92)

12. Secondary Outcome: Peak Expiratory End Pressure (PEEP)
Description: Change from baseline in PEEP, measured using mean and standard deviation.
Time Frame: Through 24 hours
Population: All participants that received study medication
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | Lyophilized Lucinactant
Number analyzed (Participants) | 19
cm H2O | -0.1 (1.66)

13. Secondary Outcome: Ventilation Index (VI)
Description: Change from baseline in VI, defined as (Respiration Rate [RR]) × (Peak Inspiratory Pressure [PIP] - Positive End Expiratory Pressure [PEEP]) × (Partial Pressure of Arterial Carbon Dioxide (PaCO2)] / (1000), measured using mean and standard deviation. The VI is used to determine the severity of respiratory illness, with higher values indicating worsening respiratory illness.
Time Frame: Baseline through 24 hours post initiation of dosing
Population: All participants that received study medication
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Lyophilized Lucinactant
Number analyzed (Participants) | 19
index | -3.75 (15.479)

14. Secondary Outcome: Lung Compliance (CL)
Description: Change from baseline in lung compliance measured using measured using mean and standard deviation.
Time Frame: Baseline through 24 hours post initiation of dosing
Population: All participants that received study medication
Measure: Mean (Standard Deviation); unit: mL/cm H2O
Arm/Group | Lyophilized Lucinactant
Number analyzed (Participants) | 19
mL/cm H2O | 9.59 (25.251)

15. Secondary Outcome: Daily Lung Compliance (Static) on Ventilator
Description: Change from baseline in daily lung compliance (static) on ventilator using measured using mean and standard deviation.
Time Frame: Baseline through 24 hours post initiation of dosing
Population: All participants that received study medication
Measure: Mean (Standard Deviation); unit: mL/cm H2O
Arm/Group | Lyophilized Lucinactant
Number analyzed (Participants) | 19
mL/cm H2O | 2.83 (14.176)

16. Secondary Outcome: Ventilator Free Days
Description: Ventilator free days measured using mean and standard deviation.
Time Frame: Baseline through 30 days post initiation of dosing
Population: All participants that received study medication
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Lyophilized Lucinactant
Number analyzed (Participants) | 19
Days | 10.3 (12.07)

17. Secondary Outcome: Days in the Intensive Care Unit (ICU)
Description: Days in the intensive care unit (ICU) measured using mean and standard deviation.
Time Frame: Baseline through 30 days post initiation of dosing
Population: All participants that received study medication
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Lyophilized Lucinactant
Number analyzed (Participants) | 19
Days | 18.6 (9.41)

18. Secondary Outcome: Days in the Hospital
Description: Days in the hospital measured using mean and standard deviation.
Time Frame: Baseline through 30 days post initiation of dosing
Population: All participants that received study medication
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Lyophilized Lucinactant
Number analyzed (Participants) | 19
Days | 21.9 (8.31)

19. Secondary Outcome: All-cause Mortality
Description: Number of participant deaths.
Time Frame: Baseline through 30 days post initiation of dosing
Population: All participants that received study medication
Measure: Count of Participants; unit: Participants
Arm/Group | Lyophilized Lucinactant
Number analyzed (Participants) | 19
Participants | 7

20. Secondary Outcome: Organ Failure Free Days
Description: Organ failure free days measured using mean and standard deviation.
Time Frame: Baseline through 30 days post initiation of dosing
Population: All participants that received study medication
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Lyophilized Lucinactant
Number analyzed (Participants) | 19
Days | 5.7 (6.44)

ADVERSE EVENTS:
Time Frame: Enrollment to 30 days after enrollment
Arm/Group | Lyophilized Lucinactant
All-Cause Mortality (participants affected / at risk) | 7/19
Serious Adverse Events (participants affected / at risk) | 8/19
Other Adverse Events (participants affected / at risk) | 16/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lyophilized Lucinactant (N=19)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) — Pneumonia as a result of COVID-19
Fungaemia (Infections and infestations) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) — Sepsis as a result of SARS-CoV-2
Septic Shock (Infections and infestations) | 2 (2)
Staphylococcal infection (Infections and infestations) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia staphylococcal (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Surgical and medical procedures (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung assist device therapy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lyophilized Lucinactant (N=19)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1)
Fungaemia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 1 (1)
Blood gases abnormal (Investigations) | 1 (1)
Oxygen saturation decreased (Investigations) | 3 (3)
Staphylococcus test positive (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia staphylococcal (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Pulmonary embolism (Vascular disorders) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Small number of subjects. No control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The preparation and submittal for publication of a manuscript containing the study results shall be in accordance with a process determined by a mutual written agreement among Windtree and participating institutions.

The publication or presentation of any study results shall comply with all applicable privacy laws, including but not limited to HIPAA. Every attempt will be made to publish results in peer-reviewed journals.

DOCUMENTS (3):
  • Study Protocol (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT04389671/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT04389671/SAP_001.pdf
  • Informed Consent Form (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT04389671/ICF_002.pdf